CLINICAL TRIAL: NCT02889263
Title: Comparison of Rehospitalization Rates in France and the United States
Acronym: REHOSP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUANTIN DGOS 2015
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Individuals Hospitalized for Any Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The problem of rehospitalizations in the US is well documented but poorly understood. Although Medicare compares the rates of rehospitalization across the country, we have found no comparison of different countries. This is a first attempt to compare rehospitalization in the US with France where national health insurance (NHI) provides easy access to primary care but, like the US, policymakers struggle to improve coordination between hospitals and community-based health care providers.Although France's NHI system with central state intervention differs from the United States' tradition of federalism, private health insurance and pluralism, policymakers seek to achieve cost savings and to reform the health care system. A recent literature review on avoidable rehospitalization of older persons in France cited studies on the topic and relied largely on ones from the US. Starting in 2013, the Center for Medicare and Medicaid Services' (CMS) 'Hospitals Readmissions Reductions Program' withheld up to 1% of regular reimbursements for hospitals with higher than expected (by CMS) rates of rehospitalization, within 30 days of discharge, due to heart attacks, heart failure and pneumonia. CMS increased this to 2% in 2014, will raise it to 3% in 2015 and may subsequently expand the list of conditions for which it will penalize early rehospitalizations. Policymakers in France have been reluctant to implement a hospital pay for performance system based on a rehospitalization indicator whose validity is a subject of considerable controversy. Despite the controversy and differences in approach, a comparison of rehospitalizations between the US and France provides a cross-national perspective on a timely policy issue facing both countries.

DETAILED DESCRIPTION:
Data sources :

The hospital administrative data for this study are from the SNIIRAM (Syste'me National d'Informations Inter Regimes de l'Assurance Maladie) which also includes the national hospital reporting system (PMSI - Programme de Medicalisation des Systemes d'Information. The SNIIRAM is a centralized administrative database of all health services reimbursed under France's NHI program. The PMSI, based on diagnosis-related groups (DRGs), is a centralized administrative database of hospital discharge records by diagnosis, procedure, age and residence of patients from all hospitals in France. It is managed by a national agency (ATIH).

To calculate the proportion of rehospitalized patients (65þ) who received outpatient visits (all physician consultations in community-based practice, as well as hospital outpatient visits) between the time of discharge and rehospitalization, we collaborated with analysts at the French NHI fund (CNAMTS). We linked the individual identifying variable for rehospitalized patients and extracted the outpatient visits from the SNIIRAM database for all medical and surgical admissions. Of the total number of hospitalized French patients aged 18 years and over (5,804,677) with identifiers in 2010, only 299,364 (5%) were unidentified after linking these datasets. These patients are most likely to have been foreigners and newborns who had not yet received an identifier. Outpatient visits include all physician consultations in community-based practice, as well as hospital outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged over 65 years in France in 2010

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients aged over 65 years in France in 2010
Sampling Method: Non-Probability Sample
Enrollment: 1944566 (Actual)
Dates: Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The total number of rehospitalizations within 30 days of discharge, as a percent of total hospital discharges for all acute-care hospitals | 30 days

SECONDARY OUTCOMES:
the most common diagnoses associated with the rehospitalizations for initial medical and surgical discharges | 30 days
regional patterns of rehospitalization | 30 days
the proportion of rehospitalized patients who received outpatient visits between the time of discharge and rehospitalization | 30 days